CLINICAL TRIAL: NCT01125917
Title: A Multicenter, Randomized, Double-blind, Active Comparator Study to Determine the Efficacy and Safety of BTDS 20 or Oxycodone Immediate-Release Vs Buprenorphine Transdermal System (BTDS) 5 in Subjects With Moderate to Severe Low Back Pain: A 52-Week Open-label Extension Phase of BUP3015
Brief Title: Safety of BTDS in Subjects With Low Back Pain: A 52-Week Extension Phase of BUP3015
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early due to administrative reasons.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP3015S
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Low back pain; Opioid; Transdermal
MeSH Terms: conditions — Low Back Pain | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTDS (Experimental): Buprenorphine transdermal patch
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear.
  Other Names: Butrans™
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 10 mcg/h applied for 7-day wear.
  Other Names: Butrans™
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear.
  Other Names: Butrans™

SUMMARY:
The purpose of the extension phase is to evaluate the long-term safety and tolerability of buprenorphine transdermal system (BTDS). Subjects begin the extension phase on BTDS 5 mcg/h and may up- or down-titrate the dose [up to BTDS 20 micrograms (mcg) / hour (h)] depending on adequate pain relief and tolerability.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed all visits of the double-blind phase on study drug, and subjects who discontinued study drug due to lack of therapeutic effect in the double-blind phase but completed all visits of the double-blind phase off study drug are eligible to enroll in the extension phase.
* For subjects entering the extension, 4 electrocardiograms (ECGs) are required at entry if none were collected prior to randomization while on BTDS 20. NOTE: Subjects with any 1 QT data corrected for heart rate using the Fridericia formula (QTcF) interval ≥ 500 milliseconds (msec) would be discontinued from the extension phase

Exclusion Criteria:

* Subjects requiring long-acting opioid analgesics [once- or twice-daily dosing with a every (q) 24 hours (h) or q12h drug] or transdermal fentanyl during the extension phase should be discontinued from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2004-06; Primary Completion 2005-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Steiner, MD, MS, Study Director — Purdue Pharma LP
Locations (84):
- United States (84):
  - Birmingham Pain Center, Birmingham, Alabama
  - Arthritis Clinical Intervention Program, Birmingham, Alabama
  - Winston Physician Services, Inc, Haleyville, Alabama
  - Arizona Research Center Inc, Phoenix, Arizona
  - Radiant Research, Phoenix, Arizona
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Hot Springs Pain Clinic, Hot Springs, Arkansas
  - NuLife Clinical Research, Inc., Anaheim, California
  - Lovelace Scientific Resources, Beverly Hills, California
  - Northern California Research Corp, Carmichael, California
  - International Clinical Research Network, Chula Vista, California
  - Shreenath Clinical Service, Fountain Valley, California
  - U of Calif at Davis, Med Ctr, Pain Management Center, Sacramento, California
  - Accelovance, San Diego, California
  - Southern Colorado Clinic, Pueblo, Colorado
  - Chiefland Medical Center, Chiefland, Florida
  - University Clinical Research Deland, DeLand, Florida
  - Drug Study Institute, Jupiter, Florida
  - Innovative Research of West Florida, Inc., Largo, Florida
  - Renstar Medical, Ocala, Florida
  - Peninsula Research Inc., Ormond Beach, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Georgia Medical Research Institute, Marietta, Georgia
  - Atlanta Knee & Shoulder Clinic, Stockbridge, Georgia
  - Pain Care Boise, Boise, Idaho
  - Idaho Arthritis and Osteoporosis Center, Meridian, Idaho
  - Pain and Rehabilitation Clinic of Chicago, Chicago, Illinois
  - GFI Research Center, Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Medical Associates Clinics, Dubuque, Iowa
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - CTT, Inc., Prairie Village, Kansas
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - New Orleans Clinical Trial Management Inc., Metairie, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - Research Center of Louisiana, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Future Care Studies, Springfield, Massachusetts
  - Rheumatology PC, Kalamazoo, Michigan
  - Lake Michigan Clinical Research & Consulting, Inc., Saint Joseph, Michigan
  - Medex Healthcare Research Inc, St Louis, Missouri
  - HealthCare Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Lovelace Scientific Resources, Henderson, Nevada
  - Pivotal Research Centers, North Las Vegas, Nevada
  - Research Across America, New York, New York
  - Pain and Orthopedic Neurology , Charlotte Spine Center,, Charlotte, North Carolina
  - Metrolina Medical Research, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, Durham, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - MedArk Clinical Research, Morgantown, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Odyssey Research, Bismarck, North Dakota
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Associated Medical Services Inc, Oklahoma City, Oklahoma
  - Keystone Clinical Research, Altoona, Pennsylvania
  - Valley Pain Specialists, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Central Pennsylvania Clinical Research, Mechanicsburg, Pennsylvania
  - BioMedical Research Associates, Shippensburg, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - New England Center Clinical Research, Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - The Arthritis and Osteoporosis Center, Orangeburg, South Carolina
  - Brown Clinic, Watertown, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - Tri Cities Medical Research, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Galenos Research, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Team Research of Central Texas, Harker Heights, Texas
  - KRK Medical Research, Richardson, Texas
  - Benchmark Research, San Angelo, Texas
  - Unlimited Research, San Antonio, Texas
  - Texas Medical Research Associates, San Antonio, Texas
  - Clinical Trial Network Oaks Medical Center, Spring, Texas
  - N. Texas Neuro Research, Wichita Falls, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Dean Medical Center, Oregon, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study dates: 17-Jun-2004 to 23-Sep-2005 at 52 medical/research sites in the United States participated in the extension study.
Pre-assignment Details: Subjects who completed all visits of the 12-week double-blind phase on study drug as well as subjects who both discontinued study drug due to lack of therapeutic effect in the double-blind phase and completed all visits of the double-blind phase off study drug were eligible for enrollment in the extension phase.
Groups:
- Total BTDS 5, 10, 20: Test treatment: Open-label buprenorphine transdermal patch 5, 10, or 20 mcg/h applied for 7-day wear
Period: Overall Study
Arm/Group | Total BTDS 5, 10, 20
Started | 354
Completed | 15
Not Completed | 339
Not completed — Adverse Event | 43
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 31
Not completed — Administrative | 223
Not completed — Lack of Efficacy | 19

BASELINE CHARACTERISTICS:
Arm/Group | Total BTDS 5, 10, 20
Number analyzed (Participants) | 354
Age Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 197

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety
Description: The purpose of the extension phase was to evaluate the long-term safety and tolerability of BTDS in subjects who had participated in the core study (BUP3015).
Time Frame: 52-week extension phase
Population: The Extension Safety Population (N = 354) consisted of all subjects who received at least 1 dose of the open-label BTDS extension study drug, and had at least 1 safety assessment during the extension phase.
Measure: Number; unit: participants
Arm/Group | Total BTDS 5, 10, 20
Number analyzed (Participants) | 354
participants
  Death | 1
  Serious adverse events | 20
  All other adverse events in ≥ 4.5% of subjects | 153

ADVERSE EVENTS:
Time Frame: Adverse events(AEs) that occurred after the signing of the informed consent up to end of study and 7 days after, discontinuation, or serious AEs occurring up to 30 days following the last study visit were followed until the AE or sequelae resolved.
Description: AEs were learned of by spontaneous reports, subject interview, and daily diary.
Arm/Group | Total BTDS 5, 10, 20
Serious Adverse Events (participants affected / at risk) | 20/354
Other Adverse Events (participants affected / at risk) | 153/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total BTDS 5, 10, 20 (N=354)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Intractable nausea (Gastrointestinal disorders) | 1 (2)
Intractable vomiting (Gastrointestinal disorders) | 1 (2)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Acute cardiac death (General disorders) | 1 (1) — DEATH
Angina (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Chest pressure (General disorders) | 1 (1)
Acalculous cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Helicobacter pylori (Infections and infestations) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Implant failure left knee (Injury, poisoning and procedural complications) | 1 (1)
Spinal column blood clot secondary to T11-12 laparoscopic cyst removal (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Acute mid back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative joint disease, right hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening of left knee OA (Musculoskeletal and connective tissue disorders) | 1 (1)
Sigmoid colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Probable seizure disorder (Nervous system disorders) | 1 (1)
Progression of lumbar spinal stenosis (Nervous system disorders) | 1 (1)
Acute exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cocaine abuse (Social circumstances) | 1 (1)
Placental abruption (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Poststudy SAE. Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total BTDS 5, 10, 20 (N=354)
Nausea (Gastrointestinal disorders) | 34
Application site pruritus (General disorders) | 37
Application site erythema (General disorders) | 36
Application site rash (General disorders) | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 27
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 16
Headache (Nervous system disorders) | 55

LIMITATIONS AND CAVEATS:
BUP3015S was terminated early due to administrative reasons unrelated to efficacy or safety. There was full evaluation of safety but no evaluation of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days